CLINICAL TRIAL: NCT00201344
Title: A Phase III Study of Radiotherapy With or Without Adjuvant Chemotherapy in Advanced Stage Nasopharyngeal Carcinoma Patients
Brief Title: A Phase III Study of Radiotherapy With or Without Adjuvant C/T in Advanced Stage Nasopharyngeal Carcinoma Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); Kaohsiung Medical University (Other); Kaohsiung Veterans General Hospital. (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1394
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2009-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Radiotherapy; Adjuvant chemotherapy; Chemtherapy; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

INTERVENTIONS:
Drug: Cisplatin,5-FU,Leucovorin

SUMMARY:
* To investigate the efficacy of adjuvant PFL chemotherapy after radiotherapy vs radiotherapy alone in AJC stage IV nasopharyngeal carcinoma patients. The endpoints of the study includes : overall survival, relapse free survival, distant metastasis and local-regional control rates.
* To evaluate the toxicities of the two treatment methods.

DETAILED DESCRIPTION:
The head and neck contracts study tested induction and maintenance chemotherapy in patients with advanced head and neck cancers.There were no significant differences in survival between the two groups, but disease free survival was prolonged in the maintenance arm and not in the induction arm. Time to and frequency of distant metastases as the first site of relapse were significantly better for those on the maintenance arm. Many trials, designed several years ago, delivered single agent chemotherapy and were not particularly intensive. Most clinical trials were dealing with a heterogenous group of head and neck cancer patients. We felt that a better choice of adjuvant chemotherapy on cancers should include: (1) localized cancers with high metastatic potential following effective local treatment; (2) effective chemotherapy available; (3) chemotherapy should be intensive and effective enough to avoid the development of drug resistance. Of course, NPC had long been regarded as one of the most suitable head and neck cancers that may benefit from adjuvant chemotherapy due to its unique high response rate to chemotherapy and high metastatic potential after radiotherapy for localized, advanced staged disease.

If radiotherapy plus adjuvant chemotherapy can improve the treatment results of standard radiotherapy by increasing the survival rate, decreasing the metastatic rate and local recurrence rate, then many NPC patients may benefit.

Therefore, we propose this phase III study of radiotherapy with or without adjuvant PFL chemotherapy in advanced stage NPC patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven nasopharyngeal carcinoma who have just completed curative radiotherapy treatment.
* Original stage must be stage IV disease (M0)
* Patients must have a complete response, partial response or stable disease assessed 4 weeks after radiotherapy.
* Performance status scale ECOG grade 0，1.
* Creatinine ≦ 1.5mg/dl and bilirubin ≦ 2.0mg/dl, WBC ≧ 3,000/mm3 and PLT ≧ 100,000/mm3,or Creatinine Clearance > 45ml/min if Creatinine > 1.5mg/dl.
* Patients must be younger than 70 year-old.
* Patients must give signed informed consent.

Exclusion Criteria:

* Patients had progressive disease after radiotherapy
* Patients had evidence of distant metastasis.
* Patients had completed radiotherapy for more than 7 weeks.
* The presence of life-threatening illness
* History of prior malignancy excluding basal cell carcinoma or squamous carcinoma of the skin or in-situ cervical cancer within 3 years of the diagnosis of NPC cancer.
* Previous chemotherapy.
* Pregnancy.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320
Dates: Start 1994-11; Study Completion 2000-01

PRIMARY OUTCOMES:
overall survival, relapse free survival,distant metastasis and local-regional control rates.

SECONDARY OUTCOMES:
toxicities of the two treatment methods.

CONTACTS AND LOCATIONS:
Overall Officials: Kwan-Hwa Chi, MD,, Principal Investigator — Taiwan cooperative oncology group
Locations (1):
- Veterans General Hospital-Taipei, Taipei, Taiwan